CLINICAL TRIAL: NCT02786732
Title: Phase 3 Study to Evaluate the Efficacy and Safety of Induction and Maintenance Regimens of Brodalumab Compared With Placebo and Ustekinumab in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Study to Evaluate Broadlumab vs Placebo and Ustekinumab
Acronym: AMAGINE-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor
Sponsor: MedDerm Associates (Industry)
Responsible Party: Principal Investigator, Michelle Pelle, M.D., Principal Investigator, MedDerm Associates
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120104
Record Dates: First submitted 2014-06-23; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab; Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 210mg Brodalumab (Experimental): Administered by subcutaneous injection until Week 12
  Interventions: Biological: 210mg Brodalumab
- 140mg Brodalumab (Experimental): Administered subcutaneous injection until Week 12
  Interventions: Biological: 210mg Brodalumab
- Ustekinumab (Active Comparator): Administered subcutaneous injection until Week 52
  Interventions: Biological: 140mg Brodalumab
- Placebo (Placebo Comparator): Administered subcutaneous injection until Week 12
  Interventions: Biological: 210mg Brodalumab; Biological: Ustekinumab; Biological: Placebo

INTERVENTIONS:
Biological: 210mg Brodalumab — Brodalumab 210mg administered subcutaneously
  Arms: 140mg Brodalumab; 210mg Brodalumab; Placebo
Biological: 140mg Brodalumab — Brodalumab 140mg administered subcutaneously
  Arms: Ustekinumab
Biological: Ustekinumab — Ustekinumab 45mg or 90mg adminstered subcutaneously
  Arms: Placebo
Biological: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Induction and Maintenance Regimens of Brodalumab compared with Placebo and Ustekinumab in subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
The study is up to 5 years. If you qualify, you will be randomized into 1 of 4 groups. Two groups will get brodalumab(1 group will get 210milligrams of brodalumab at each dose and the other group will get 140 milligrams of brodalumab at each dose), one group will get ustekinumab, and one group will get placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months before first dose of IP.
* Subject has involved body surface area >_10%, PASI>_, and sPGA>_3 at screening and at baseline.
* For women, a negative serum pregnancy test during screening a negative urine pregnancy test at baseline.
* Subject has no known history of active tuberculosis.
* Subject has a negative test for tuberculosis during screening.

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions at the time of the screening visit that would interfere with evaluations of the effect of IP on psoriasis.
* Subject has a planned surgical intervention between baseline and the week 52 evaluation.
* Subject an active infection or history of infections.
* Subject has any systemic disease considered by the investigator to be clinically significant and uncontrolled.
* Subject has known history of Crohn's disease.
* Subject has known history of hepatitis B, hepatitis C, or human immunodeficiency virus.
* Subject had myocardial infarction or unstable angina pectoris within the past 12 months prior to the first dose of IP.
* Subject has any active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma.
* Subject has history of malignancy within 5 years EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, in situ cervical cancer, or in situ breast ductal carcinoma.
* Subject has received live vaccine(s) within 28 days of the first dose of IP.
* Subject has used ustekinumab and/or antio-IL-17 biologic therapy ever or other experimental or commercially available biologi immune modulator(s) within 12weeks prior to the first IP dose
* Subject currently is enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s).
* For women not willing to use highly effective methods of birth control during treatment and for 15 weeks after the last dose.
* For women; pregnant or breast feeding, or planning to become pregnant while enrolled in the study and for 15 weeks after the last dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
PASI Improvement | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michelle T Pelle, M.D., Principal Investigator — MedDerm Associates
Locations (1):
- MedDerm Associates, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No